CLINICAL TRIAL: NCT03934684
Title: Post-marketing Phase 4 Study to Evaluate Safety, Tolerability, and Efficacy of Kyprolis® (Carfilzomib) in Indian Patients With Relapsed or Refractory Multiple Myeloma: A Prospective, Open-label, Non-comparative, Multicenter Study
Brief Title: Study to Evaluate Safety Tolerability & Efficacy of Kyprolis (Carfilzomib) in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160372
Record Dates: First submitted 2019-04-16; First posted 2019-05-02 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Relapsed Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Carfilzomib + Dexamethasone (Experimental): Drug: Carfilzomib + Dexamethasone
  * Carfilzomib 20 mg/m2 on days 1 and 2, and if tolerated, escalated to a target dose of 56 mg/m2 starting on day 8 of cycle 1 and thereafter.
  * Dexamethasone 20 mg taken by mouth or intravenously on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle. An individual subject will receive study treatment for a maximum of 3 years if the subject has not yet experienced disease progression
  Interventions: Drug: Drug: Carfilzomib + Dexamethasone
- Carfilzomib+Lenalidomide+Dexamethasone (Experimental): Drug: Carfilzomib + Lenalidomide + Dexamethasone
  * Carfilzomib is 20 mg/m2 on days 1 and 2, and if tolerated, escalated to a target dose of 27 mg/m2 starting on day 8 of cycle 1 and thereafter. From cycle 13, the day 8 and day 9 doses of Carfilzomib will be omitted.
  * Lenalidomide 25 mg is taken orally on days 1 to 21.
  * Dexamethasone 40 mg on days 1, 8, 15, and 22 of the 28-day cycles. An individual subject will receive study treatment for a maximum of 18 months consistent with the approved use in this combination.
  Interventions: Drug: Drug: Carfilzomib + Lenalidomide + Dexamethasone

INTERVENTIONS:
Drug: Drug: Carfilzomib + Dexamethasone — Drug: Carfilzomib + Dexamethasone
  * Carfilzomib will be administered as a 30-minute infusion.
  * Dexamethasone will be taken by mouth or intravenously.
  Other Names: Kyprolis
  Arms: Carfilzomib + Dexamethasone
Drug: Drug: Carfilzomib + Lenalidomide + Dexamethasone — Drug: Carfilzomib + Lenalidomide + Dexamethasone
  * Carfilzomib will be administered as a 10 minute infusion.
  * Lenalidomide will be taken orally.
  * Dexamethasone will be taken by mouth or intravenously.
  Other Names: Kyprolis
  Arms: Carfilzomib+Lenalidomide+Dexamethasone

SUMMARY:
To characterize safety associated with the use of Kyprolis under the locally approved label.

DETAILED DESCRIPTION:
Kyprolis® (K; carfilzomib) was approved in India on 17 January 2017 as a prescription medication in combination with dexamethasone (Kd) or with lenalidomide (Revlimid®) plus dexamethasone (KRd) for the treatment of patients with relapsed or refractory multiple myeloma (RRMM) following 1 to 3 prior lines of therapy.

This non-comparative, interventional phase 4 study is designed to fulfil the post-marketing requirement to assess safety, tolerability, and efficacy of Kyprolis on Indian subjects with RRMM as per the locally approved label.

ELIGIBILITY:
Inclusion Criteria:

* Documented RRMM after last treatment. Refractory is defined as meeting 1 or more of the following: Nonresponsive to most recent therapy (stable disease [SD] or progressive disease [PD]) while on treatment, or Disease progression within 60 days of discontinuation from the most recent therapy.
* Eligible to receive Kyprolis per the locally approved label.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Adequate hepatic function within 28 days prior to enrollment: bilirubin < 1.5 times the upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times the ULN.
* Absolute neutrophil count (ANC) ≥ 1.0 x 10^9 /L within 28 days prior to enrollment. (Screening ANC should be independent of granulocyte- and granulocyte macrophage-colony stimulating factor support for at least 1 week and of pegylated granulocyte stimulating factor for ≥ 2 weeks).
* Hemoglobin ≥ 80 g/L within 28 days prior to enrollment. Subjects should not have received red blood cell (RBC) transfusions for at least 7 days prior to obtaining the screening hemoglobin.
* Platelet count ≥ 75 x 10^9/L (≥ 50 x 10^9/L if myeloma involvement in the bone marrow is ≥ 50%) within 28 days prior to enrollment. Subjects should not have received platelet transfusions for at least 7 days prior to obtaining the screening platelet count.
* Adequate renal function within 28 days prior to enrollment (either measured or calculated using a standard formula such as the Cockcroft and Gault): calculated or measured creatinine clearance (CrCl) of ≥ 50 mL/min for subjects receiving KRd; calculated or measured CrCl of ≥ 15 mL/min for subjects receiving Kd.
* Left ventricular ejection fraction ≥ 40% as assessed by transthoracic echocardiogram (TTE) or multigated acquisition scan (MUGA).
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test within the 10 to 14 days prior to enrollment and a negative urine pregnancy test within the 24 hours prior to day 1 of each cycle prior to dosing.
* Subject or legally acceptable representative has provided informed consent/assent prior to initiation of any study specific activities/procedures.

Exclusion Criteria:

* Waldenström macroglobulinemia.
* Plasma cell leukemia (> 2.0 x 10^9/L circulating plasma cells by standard differentials).
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Myelodysplastic síndrome.
* Primary amyloidosis (subjects with multiple myeloma with asymptomatic deposition of amyloid plaques found on biopsy would be eligible if all other criteria are met).
* History of other malignancy within the past 5 years, with the following exception[s]: Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease. Adequately treated cervical carcinoma in situ without evidence of disease. Adequately treated breast ductal carcinoma in situ without evidence of disease. Prostatic intraepithelial neoplasia without evidence of prostate cáncer. Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* Known immediate or delayed hypersensitivity reaction to Captisol (a cyclodextrin derivative used to solubilize Kyprolis).
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs.
* Intolerance to hydration.
* Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, uncontrolled arrhythmias, clinically significant echocardiogram (ECHO) abnormalities, screening ECG with corrected QT interval (QTc) of > 470 msec, pericardial disease, or myocardial infarction within 4 months prior to enrollment.
* Infiltrative pulmonary disease and/or known pulmonary hypertension.
* Active infection within 14 days prior to enrollment requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents. Such infections must be fully resolved prior to initiating study treatment.
* Pleural effusions requiring thoracentesis within 14 days prior to enrollment.
* Ascites requiring paracentesis within 14 days prior to enrollment.
* Uncontrolled hypertension, defined as an average systolic blood pressure > 159 mmHg or diastolic > 99 mm/Hg despite optimal treatment (measured following European Society of Hypertension/European Society of Cardiology [ESH/ESC] 2013 guidelines.
* Active hepatitis B virus (HBV) infection. Subjects with positive hepatitis B surface antigen (HBsAg) or core antibody (anti-HBc) that achieve sustained virologic response with antiviral therapy directed at hepatitis B are allowed. Subjects with known history or resolved infection (negative for HBsAg but positive for antibodies to surface antigen, and/or core antigen) must be screened with HBV DNA levels. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (hepatitis B surface antibody [anti-HBs] positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA.
* Known human immunodeficiency virus (HIV) infection, hepatitis C infection (subjects with hepatitis C that achieve a sustained virologic response following antiviral therapy are allowed).
* Ongoing graft-versus-host disease.
* Subjects with grade 3 or worse neuropathy within 14 days prior to enrollment.
* Antitumor therapy (eg, chemotherapy, immunotherapy, antibody therapy) or investigational agent within 28 days before enrollment or not recovered from any acute toxicity.
* Subjects on immunosuppressive therapy for graft versus host disease, even if it has resolved.
* Glucocorticoid therapy within 14 days before first dose that exceeds a cumulative dose of 160 mg or dexamethasone or equivalent dose of other corticosteroids.
* Focal radiation therapy within 7 days before enrollment. Radiation therapy to an extended field involving significant volume of bone marrow within 28 days prior to enrollment (ie, prior radiation must have been to less than 30% of the bone marrow).
* Autologous stem cell transplant less than 100 days prior to enrollment.
* Prior treatment with Kyprolis (carfilzomib).
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study. Other investigational procedures while participating in this study are excluded.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment, during any breaks (interruptions) in the treatment, and for an additional 30 days after the last dose of Kyprolis. Females of childbearing potential should only be included in the study after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test.
* Female subjects of childbearing potential unwilling to use 1 highly effective method of contraception during treatment, during any breaks (interruptions) in the treatment, and for an additional 30 days after the last dose of Kyprolis.

NOTE: Female subjects of childbearing potential being treated with lenalidomide must agree to use 2 methods of contraception for at least 28 days before starting treatment, during treatment, during any breaks (interruptions) in the treatment, and for an additional 30 days after the last dose of treatment.

• Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 90 days after the last dose of Kyprolis.

NOTE: Male subjects being treated with lenalidomide must agree to use a male condom with spermicide even if they have undergone a successful vasectomy.

* Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 90 days after the last dose of Kyprolis.
* Male subjects unwilling to abstain from donating sperm during treatment and for an additional 90 days after the last dose of Kyprolis.
* Subject likely to not be available to complete all protocol required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Active hepatitis B virus (HBV) infection. Subjects with positive hepatitis B surface antigen (HBsAg) or core antibody (anti-HBc) that achieve sustained virologic response with antiviral therapy directed at hepatitis B are allowed. Subjects with known history or resolved infection (negative for HBsAg but positive for antibodies to surface antigen, and/or core antigen) must be screened with HBV DNA levels. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (hepatitis B surface antibody [anti-HBs] positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2025-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- India (17):
  - Yashoda Hospital, Hyderabad, Andhra Pradesh
  - Apollo Hospital, Hyderabad, Andhra Pradesh
  - M S Ramaiah Memorial Hospital, Bangalore, Karnataka
  - K L E S Dr Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - Cytecare Cancer Hospitals, Bengaluru, Karnataka
  - Aster Medcity, Kochi, Kerala
  - Government Medical College, Kozhikode, Kerala
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Mumbai Oncocare Center, Mumbai, Maharashtra
  - Navsanjeevani Hospital, Nashik, Maharashtra
  - Heath Care Group Manavata Cancer Centre, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, Puducherry
  - Cancer Institute WIA, Chennai, Tamil Nadu
  - Thangam Cancer Centre, Namakkal, Tamil Nadu
  - Valentis Cancer Hospital, Meerut, Uttar Pradesh
  - Netaji Subhash Chandra Bose Cancer Research Institute, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 101 participants were enrolled into this study at 15 centers in India. The analyses presented in this results summary are based on the primary completion data. The primary completion data cut-off was 23 March 2023. The study is ongoing.
Pre-assignment Details: Screening assessments were conducted within 28 days before enrollment into the study.
Groups:
- Carfilzomib, Lenalidomide and Dexamethasone (KRd): Participants with relapsed or refractory multiple myeloma received a triplet combination of KRd.
  Carfilzomib was administered as a 10-minute intravenous (IV) infusion on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day treatment cycles. The starting dose of carfilzomib was 20 mg/m^2 on Days 1 and 2, and if tolerated, escalated to a target dose of 27 mg/m^2 starting on Day 8 of cycle 1 and thereafter. From cycle 13, the Day 8 and Day 9 doses of carfilzomib were omitted. After cycle 18, carfilzomib was discontinued.
  Lenalidomide 25 mg was taken orally on Days 1 to 21 and dexamethasone 40 mg by mouth or IV infusion on Days 1, 8, 15, and 22 of repeated 28-day treatment cycles.
- Carfilzomib and Dexamethasone (Kd): Participants with relapsed or refractory multiple myeloma received a doublet combination of Kd.
  Carfilzomib was administered as a 30-minute IV infusion on Days 1, 2, 8, 9, 15, and 16 of repeated 28-day treatment cycles. The starting dose of carfilzomib was 20 mg/m^2 on Days 1 and 2, and if tolerated, was escalated to a target dose of 56 mg/m^2 starting on Day 8 of cycle 1 and thereafter.
  Dexamethasone 20 mg was taken by mouth or intravenously on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle.
Period: Overall Study
Arm/Group | Carfilzomib, Lenalidomide and Dexamethasone (KRd) | Carfilzomib and Dexamethasone (Kd)
Started | 49 | 52
Completed | 7 | 3
Not Completed | 42 | 49
Not completed — Participants continuing in study | 11 | 4
Not completed — Discontinuation of carfilzomib | 20 | 30
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 7 | 8

BASELINE CHARACTERISTICS:
Population: Measured in the full analysis set, which included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Carfilzomib, Lenalidomide and Dexamethasone (KRd) | Carfilzomib and Dexamethasone (Kd) | Total
Number analyzed (Participants) | 49 | 52 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (8.2) | 61.9 (9.9) | 59.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 32 | 37 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 52 | 101
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 52 | 101
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment(s). TEAEs were graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.4.03. Any clinically significant laboratory changes over time were recorded as TEAEs.
Time Frame: From the first dose date of any study drug until the end of study or cutoff date, whichever occurred earlier (median [min, max] time on treatment was 43.14 [4.4, 73.4] weeks for the KRd group and 28.79 [0.3, 107.3] weeks for the Kd group)
Population: Measured in the safety analysis set, which included all enrolled participants who received at least one dose of the investigational product(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib, Lenalidomide and Dexamethasone (KRd) | Carfilzomib and Dexamethasone (Kd)
Number analyzed (Participants) | 49 | 52
Participants | 46 | 43

2. Primary Outcome: Number of Participants Who Experienced Serious TEAEs
Description: A serious TEAE is any untoward medical occurrence in a clinical study participant after first dose irrespective of a causal relationship with the study treatment(s) that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib, Lenalidomide and Dexamethasone (KRd) | Carfilzomib and Dexamethasone (Kd)
Number analyzed (Participants) | 49 | 52
Participants | 12 | 19

ADVERSE EVENTS:
Time Frame: For all-cause mortality reporting, from enrollment until the end of study, death date or cutoff date, whichever occurred earlier (median [min, max] time on study was 8.7 [0.1, 25.6] months). For serious and other adverse event reporting, from the first dose date of any study drug until the end of study or cutoff date, whichever occurred earlier (median [min, max] time on treatment was 43.14 [4.4, 73.4] weeks for the KRd group and 28.79 [0.3, 107.3] weeks for the Kd group)
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Carfilzomib, Lenalidomide and Dexamethasone (KRd) | Carfilzomib and Dexamethasone (Kd)
All-Cause Mortality (participants affected / at risk) | 2/49 | 2/52
Serious Adverse Events (participants affected / at risk) | 12/49 | 19/52
Other Adverse Events (participants affected / at risk) | 45/49 | 41/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib, Lenalidomide and Dexamethasone (KRd) (N=49) | Carfilzomib and Dexamethasone (Kd) (N=52)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Acute cardiac event (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiotoxicity (Cardiac disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia acinetobacter (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib, Lenalidomide and Dexamethasone (KRd) (N=49) | Carfilzomib and Dexamethasone (Kd) (N=52)
Anaemia (Blood and lymphatic system disorders) | 7 | 18
Leukopenia (Blood and lymphatic system disorders) | 5 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 7 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 12
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 11
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 5 | 9
Fatigue (General disorders) | 3 | 9
Oedema peripheral (General disorders) | 4 | 3
Pyrexia (General disorders) | 8 | 13
Cellulitis (Infections and infestations) | 0 | 4
Lower respiratory tract infection (Infections and infestations) | 4 | 1
Nasopharyngitis (Infections and infestations) | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Headache (Nervous system disorders) | 0 | 5
Hypoaesthesia (Nervous system disorders) | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 6
Paraesthesia (Nervous system disorders) | 4 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT03934684/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03934684/SAP_001.pdf